CLINICAL TRIAL: NCT02803086
Title: Longitudinal Evaluation of Intestinal, Haematological and Urinary Toxicity From Pelvic Irradiation for Prostate Cancer
Acronym: IHU-WPRT-TOX
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Regina Elena Cancer Institute (Other); Azienda Ospedaliero Universitaria, Santa Maria della Misericordia di Udine, Italy (Other); Cliniche Humanitas Gavazzeni (Other); Centro AKTIS Diagnostica e Terapia (Unknown); Azienda Sanitaria dell'Alto Adige (Other); Azienda Sanitaria Locale To4 (Unknown); Azienda USL Reggio Emilia - IRCCS (Other Government); Candiolo Cancer Institute - IRCCS (Other); Azienda Sanitaria Locale di Biella (Other); Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other); Azienda U.S.L. della Valle d'Aosta (Unknown); IRCCS Centro di Riferimento Oncologico della Basilicata (Other)
Responsible Party: Principal Investigator, Cesare Cozzarini, MD, IRCCS San Raffaele
Other Study IDs: IRCCS San Raffaele
Record Dates: First submitted 2016-06-08; First posted 2016-06-16 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Radiotherapy; Hematopoietic stem cells; Radiotoxicity
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: To date, around 700 patients, who were treated with Radiotherapy for Prostate Cancer, have been enrolled. 34% of them underwent radiotherapy with radical intent, whereas the others were post-prostatectomy patients (29% adjuvant, 37% salvage). Various techniques of irradiation were used (1% 3DCRT, 6% SF-IMRT, 52% VMAT, 41% Tomotherapy) in conventional (42%, 1.7-2.0 Gy/fr.) and hypofractionated (58%, 2.1-2.7 Gy/fr.) settings. EQD2(alpha/beta=3) to prescribed PTV ranged between 64 and 93 Gy. Limph nodes were treated in the 98% of cases.

SUMMARY:
The prophylactic irradiation of pelvic lymph-nodes by means of Whole-Pelvis Radiotherapy (WPRT) in the treatment of prostate cancer (PCa) is aimed at the timely eradication of microscopic lymph-nodal metastases. Nevertheless, even though delivered by means of modern Intensity-Modulated Radiotherapy (IMRT) techniques, WPRT may result in intestinal, hematologic and urinary toxicity (IT, HT, UT, respectively) severely affecting patients' daily health-related quality-of-life (HRQoL) within the so-called and inadequately investigated Pelvic Radiation Disease.

The aim of this study is to develop sophisticated predictive models of IMRT-WPRT induced patient-reported HT, IT and UT in PCa. The possible correlation between several clinical factors and radiation doses received by various pelvic structures (i.e. pelvic bones subvolumes, intestinal loops, sigmoid, rectum and bladder) and risk and severity of patient-reported IT, UT and HT will be analyzed and robust multi-variable models will be developed and internally validated. A secondary end-point will be the identification of specific symptoms affecting patients' HRQoL during irradiation and in the long term, overall and in different therapeutic settings (radical, adjuvant and salvage). Lastly, possible correlation between HT and UT/IT will be investigated.

DETAILED DESCRIPTION:
Experimental Design:

Hypothesis. Dose-volume histograms (DVHs) of bowel, sigmoid colon and rectum are expected to be predictive of IT prospectively self-assessed by patients by means of IBDQ (Inflammatory Bowel Disease Questionnaire). Similarly, DVHs of pelvic bony subvolumes (lumbar-sacral, iliac and the lower pelvis) should predict HT, while DVHs and dose-surface histograms (DSHs) of the bladder are expected to be predictive of UT self-assessed by patients by means of IPSS (International Prostate Symptoms Score) and ICIQ-SF (International Consultation on Incontinence Questionnaire- short form) questionnaires. Moreover, some specific urinary and intestinal-rectal symptoms are expected to lead to impairment in emotional, social and systemic domains, as assessed by the IBDQ questionnaire, more than others, with several possible "clusters" of symptoms prevailing in different treatment settings. Finally, the intestinal, urinary and hematologic toxicity profile of WPRT IMRT could emerge to be extremely different in patients treated with radical (RAD), adjuvant (ADV) or salvage (SALV) intent.

Task1. The principal aim of the project is to develop sophisticated quantitative predictive models of IT, UT and HT (without the confounding bias of chemotherapy) from WPRT IMRT in both radical and postoperative treatment of localized PCa. The possible correlation between the radiation doses received by different pelvic structures and different toxicities will be analyzed.

Task2. To try to individuate the intestinal/rectal and urinary symptoms most negatively affecting the Emotional, Social and Systemic patient domains, with the ultimate objective of "focusing" the quantitative predictive models including both clinical and physico-dosimetric parameters only upon these main symptoms. This approach could theoretically permit the creation of a "shortened and radiotherapy adapted" version of the IBDQ questionnaire.

Task3. A thorough assessment of the different self-assessed toxicity profiles to be expected in patients treated with RAD, ADV or SALV intent will be carried out, with the ultimate aim of accumulating a set of extremely detailed information to be provided to patients in order to offer them appropriate counselling after the initial diagnosis of PCa with regard to the choice between radiotherapy vs surgery. In those selecting the latter and in the presence of risk factors at prostatectomy suggesting a possible role for postoperative radiotherapy, the ultimate objective would be that of assisting patients in the always extremely problematic choice between immediate adjuvant and timely, postponed, salvage irradiation in the case of biochemical recurrence.

Task4. Secondary end-points: to search for a possible correlation between HT and IT/UT.

Throughout the treatment period, patients will be seen every 2 weeks for toxicity monitoring. Subsequently, a follow-up visit will be performed at 3 months from the end of treatment, and every six months thereafter, up to 5 years.

Intestinal and urinary toxicities, including urinary incontinence, will be self-assessed by patients by means of the Italian validated version of the IBDQ, IPSS and ICIQ-SF questionnaires: at baseline (no more than 30 days before RT start), at radiotherapy mid-point and end, at 3, 6,12, 18, 24, 30, 36, 42, 48, 54 and 60 months from radiotherapy conclusion.

A blood sample for white blood cells (WBC), with absolute neutrophil and lymphocyte counts (ANC and ALC, respectively), red blood cells (RBC) and platelets (PLT) counts will be collected at the same time intervals. In addition to the self-reported assessment of rectal/bowel and urinary symptoms during and after radiotherapy, an evaluation of acute and late IT and UT will be performed by the medical staff for possible future comparison between its subjective and objective measurement. IT, HT and UT will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.03.

ELIGIBILITY:
Inclusion Criteria:

* Patients with with an ECOG PS 0-1
* Patients with histologically proven adenocarcinoma of the prostate
* WPRT can be delivered with both static and rotational IMRT techniques such as volumetric modulated arc therapy (VMAT) or Tomotherapy
* Both conventionally (1.8-2 Gy/fraction) and moderately hypo-fractionated (≤ 2.7 Gy/fraction) regimens with simultaneous integrated boost (SIB) approach are allowed; in any case the daily dose delivered to the pelvic nodes should be in the range of 1.8-2.0 Gy/fr

Exclusion Criteria:

* Patients older than 80 years at the time of enrollment
* Missing written informed consent

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven adenocarcinoma of the prostate, candidate to radical or postoperative (both adjuvant and salvage) radiotherapy including prophylactic irradiation of the pelvic lymph-nodal area. The indication for WPRT will be at the discretion of the referring Radiation Oncologist.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2014-02; Primary Completion 2021-12 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hematologic toxicity | 5 years
  if any, acute (<within 90 days from radiotherapy completion) and late (>90 days from radiotherapy completion) Grade 1, Grade 2 and Grade 3-4 leukopenia, neutropenia, lymphopenia, erythropenia, anemia, thrombocytopenia and clinico-dosimetric factors predicting them;
Intestinal toxicity | 5 years
  a worsening of 2 points or more with respect to baseline of the 10 IBDQ items investigating the Bowel Domain (items # 1, 5, 9, 13, 17, 20, 22, 24, 26 and 29, frequency of bowel movements, liquid defecation, abdominal cramps, abdominal pain, gas passage, abdominal bloating, rectal bleeding, urge to go to bathroom even if empty intestine, accidental soiling and nausea/feeling sick, respectively) and of the three cumulative items evaluating the impact of Bowel Symptoms on the Emotional, Social and Systemic Domains.

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Cozzarini, MD, Study Chair — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sini C, Fiorino C, Perna L, Noris Chiorda B, Deantoni CL, Bianchi M, Sacco V, Briganti A, Montorsi F, Calandrino R, Di Muzio N, Cozzarini C. Dose-volume effects for pelvic bone marrow in predicting hematological toxicity in prostate cancer radiotherapy with pelvic node irradiation. Radiother Oncol. 2016 Jan;118(1):79-84. doi: 10.1016/j.radonc.2015.11.020. Epub 2015 Dec 15. PMID 26702990
- [Background] Cozzarini C, Fiorino C, Da Pozzo LF, Alongi F, Berardi G, Bolognesi A, Briganti A, Broggi S, Deli A, Guazzoni G, Perna L, Pasetti M, Salvadori G, Montorsi F, Rigatti P, Di Muzio N. Clinical factors predicting late severe urinary toxicity after postoperative radiotherapy for prostate carcinoma: a single-institute analysis of 742 patients. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):191-9. doi: 10.1016/j.ijrobp.2010.09.027. Epub 2010 Nov 23. PMID 21109361
- [Background] Cozzarini C, Noris Chiorda B, Sini C, Fiorino C, Briganti A, Montorsi F, Di Muzio N. Hematologic Toxicity in Patients Treated With Postprostatectomy Whole-Pelvis Irradiation With Different Intensity Modulated Radiation Therapy Techniques Is Not Negligible and Is Prolonged: Preliminary Results of a Longitudinal, Observational Study. Int J Radiat Oncol Biol Phys. 2016 Jun 1;95(2):690-5. doi: 10.1016/j.ijrobp.2016.01.022. Epub 2016 Jan 28. PMID 27131081
- [Background] Cozzarini C, Fiorino C, Deantoni C, Briganti A, Fodor A, La Macchia M, Noris Chiorda B, Rancoita PM, Suardi N, Zerbetto F, Calandrino R, Montorsi F, Di Muzio N. Higher-than-expected severe (Grade 3-4) late urinary toxicity after postprostatectomy hypofractionated radiotherapy: a single-institution analysis of 1176 patients. Eur Urol. 2014 Dec;66(6):1024-30. doi: 10.1016/j.eururo.2014.06.012. Epub 2014 Jun 27. PMID 24985964
- [Background] Bresolin A, Faiella A, Garibaldi E, Munoz F, Cante D, Vavassori V, Waskiewicz JM, Girelli G, Avuzzi B, Villa E, Magli A, Noris Chiorda B, Gatti M, Ferella L, Maggio A, Landoni V, Aimonetto S, Sini C, Rancati T, Sanguineti G, Valdagni R, Di Muzio N, Fiorino C, Cozzarini C. Acute patient-reported intestinal toxicity in whole pelvis IMRT for prostate cancer: Bowel dose-volume effect quantification in a multicentric cohort study. Radiother Oncol. 2021 May;158:74-82. doi: 10.1016/j.radonc.2021.02.026. Epub 2021 Feb 25. PMID 33639190
- [Background] Munoz F, Sanguineti G, Bresolin A, Cante D, Vavassori V, Waskiewicz JM, Girelli G, Avuzzi B, Garibaldi E, Faiella A, Villa E, Magli A, Noris Chiorda B, Gatti M, Rancati T, Valdagni R, Di Muzio NG, Fiorino C, Cozzarini C. Predictors of Patient-Reported Incontinence at Adjuvant/Salvage Radiotherapy after Prostatectomy: Impact of Time between Surgery and Radiotherapy. Cancers (Basel). 2021 Jun 29;13(13):3243. doi: 10.3390/cancers13133243. PMID 34209562